CLINICAL TRIAL: NCT02660684
Title: A Historically-controlled, Multi-center Study to Assess the Safety and Efficacy of Tacrolimus (Prograf Capsule, Prograf Injection) and Methotrexate Combination Therapy for Prevention of GVHD in Patients Who Received Peripheral Hematopoietic Stem Cell Transplantation From a Sibling Donor
Brief Title: Study to Assess the Safety and Efficacy of Tacrolimus (Prograf Capsule/Injection) and Methotrexate (MTX) Combination Therapy for Prevention of Graft Versus Host Disease (GVHD) in Patients Who Received Peripheral Hematopoietic Stem Cell Transplantation From a Sibling Donor
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Korea, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRG-07-11-KOR
Record Dates: First submitted 2016-01-18; First posted 2016-01-21 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Graft Versus Host Disease
Keywords: Prograf; Graft versus host disease; Hematopoietic stem cell transplantation; Prophylaxis; Peripheral hematopoietic stem cell transplantation
MeSH Terms: conditions — Graft vs Host Disease | interventions — Tacrolimus; Methotrexate; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prograf + MTX (Experimental)
  Interventions: Drug: Prograf; Drug: Methotrexate
- Cyclosporine + MTX (historical control) (Active Comparator)
  Interventions: Drug: Methotrexate; Drug: Cyclosporine

INTERVENTIONS:
Drug: Prograf — Injection or oral
  Other Names: Tacrolimus
  Arms: Prograf + MTX
Drug: Methotrexate — Injection
Drug: Cyclosporine — Injection or oral
  Arms: Cyclosporine + MTX (historical control)

SUMMARY:
The objective of this study is to assess the safety and efficacy of Tacrolimus (Prograf capsule, Prograf injection) and Methotrexate combination therapy for GVHD prophylaxis in patients who received peripheral hematopoietic stem cell transplantation from a sibling donor, and to compare with data from a historical control group that administered a conventional Cyclosporine formulation.

ELIGIBILITY:
Inclusion Criteria:

* Blood diseases for a standard risk group

  * Primary remission of AML (acute myeloid leukemia)
  * Primary remission of ALL (acute lymphocytic leukemia)
  * Secondary remission of ALL (acute lymphocytic leukemia)
  * SAA (severe aplastic anemia)
  * Chronic stage CML (chronic myeloid leukemia)
  * MDS (myelodysplastic syndrome)
  * Myeloma (multiple myeloma)
* A patient who received peripheral hematopoietic stem cell transplantation from a HLA-matched sibling donor

Exclusion Criteria:

* A patient with renal impairment (serum creatinine level ≥ 1.5mg/dl or 130μmol/l, GFR≤ 30%)
* A pregnant or breastfeeding woman
* A woman who is unwilling or unable to practice appropriate contraception during the study
* A patient who is highly likely to experience aggravation during treatment due to active tuberculosis, other hepatic disease, hypertension, heart failure, chronic obstructive respiratory disease, etc.
* A patient with hypersensitivity to tacrolimus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2008-02; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Number of occurrence sites of acute GVHD occurring within 100 days after peripheral hematopoietic stem cell transplantation from a sibling donor | Day 1 up to Day 100 post-transplant
Severity of acute GVHD occurring within 100 days after peripheral hematopoietic stem cell transplantation from a sibling donor | Day 1 up to Day 100 post-transplant
  Severity is graded according to the Seattle criteria, between 1+ ~ 4+ depending on the severity of the injury of the skin, liver and digestive system, and the overall grade is classified by including the performance change.
Number of occurrence sites of chronic GVHD occurring after 100 days after peripheral hematopoietic stem cell transplantation from a sibling donor | Day 100 up to 1 year post-transplant
Classification of chronic GVHD occurring after 100 days after peripheral hematopoietic stem cell transplantation from a sibling donor | Day 100 up to 1 year post-transplant
  Depending on the extent of occurrence, it is classified as limited (present only locally) and extensive (systemic lesions). Depending on the presence of preceding acute GVHD, it is classified as progressive for a patient with preceding acute GVHD (chronic GVHD following the occurrence of acute GVHD), quiescent (chronic GVHD after relief of acute GVHD symptoms) or otherwise (de novo).
Safety as assessed by adverse events | Day 1 up to 1 year post-transplant
Safety as assessed by laboratory assessments | Day 1 up to 1 year post-transplant
  Includes hematology, biochemistry and trough plasma concentration analysis

SECONDARY OUTCOMES:
Percentage of patients alive after peripheral hematopoietic stem cell transplantation from a sibling donor | Day 1 up to 1 year post-transplant
Percentage of patients alive after peripheral hematopoietic stem cell transplantation from a sibling donor in comparison with Cyclosporine in combination with MTX | Day 1 up to 1 year post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Korea, Inc.
Locations (3):
- South Korea (3):
  - Daegu, Gyeongsangnam-do
  - Hwasun-gun, Jeonranam-do
  - Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results Web site — https://www.astellasclinicalstudyresults.com/hcp/study.aspx?ID=PRG-07-11-KOR